CLINICAL TRIAL: NCT06379737
Title: Valutazione Degli Esiti a Medio-lungo Termine Della Sindrome Long Covid in Pazienti Trattati Con un Protocollo di Riabilitazione in Ambiente Termale o in Teleriabilitazione
Brief Title: Multi-systemic Rehabilitative Interventions in Long COVID-19 Patients in Two Different Settings: a Randomized Controlled Trial
Acronym: MULTI-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Padua University General Hospital (Other)
Responsible Party: Principal Investigator, Stefano Masiero, Professor, Padua University General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 359n/AO/23; MASI_CARIVARI21_01 (Other Grant/Funding Number: Fondazione Cariparo)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Long COVID
Keywords: rehabilitation; recovery; COVID-19; health resort medicine; balneotherapy
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based rehabilitation (Active Comparator): Perform home-based rehabilitation
  Interventions: Behavioral: Multi-systemic Rehabilitation
- Health resort medicine rehabilitation (Experimental): Perform Health resort medicine rehabilitation
  Interventions: Behavioral: Multi-systemic Rehabilitation

INTERVENTIONS:
Behavioral: Multi-systemic Rehabilitation — Patients in group A underwent a 5-week rehabilitation cycle with two weekly sessions, totaling 10 sessions, in a health resort setting. The patients underwent treatments at two health resort facilities located in the Euganean Basin, Veneto, Italy, equipped with pools of the same depth, size, and water type. Each session was structured into four components:
  1. thermal mineral-rich aerosol therapy (10 minutes);
  2. dryland motor, respiratory, and proprioceptive rehabilitation in the gym (30 minutes);
  3. mineral-rich aquatic aerobic, strengthening, and balance exercises (30 minutes);
  4. cognitive enhancement interventions (30 minutes). Inhalation treatments and aquatic exercises utilized thermal mineral-rich water, specifically salsobromoiodic water, naturally springing at approximately 80°C and used in pools at a temperature of around 36°C. The chemical-physical properties of the thermal mineral-rich water employed are reported in Table I.
  Patients in group B underwent a 5-week rehabilit

SUMMARY:
Objective: This study aimed to evaluate the effectiveness of a multisystem rehabilitation program for Long Covid patients in two different settings.

Design: Randomized controlled trial. Settings: Health resort and home-based. Participants: 72 Long Covid patients. Interventions: Patients were randomly assigned into two groups: Group A (n=36) received health resort intervention, and Group B (n=36) received home-based care. Both groups underwent a 5-week rehabilitation program, involving motor, respiratory, and cognitive exercises, two sessions per week.

Outcomes: Assessments were conducted before (T0) and after treatment (T1), at 3 (T2) and 6 months (T3), including respiratory and physical function, handgrip strength, fatigue, pain, quality of life, psychological function, and satisfaction.

DETAILED DESCRIPTION:
At the outpatient clinics of the Neurorehabilitation Unit of the University Hospital of Padua, 103 patients were initially assessed. Out of these patients, 72 subjects of both genders with medium-to-long-term outcomes following previous infection with the SARS-CoV-2 virus were recruited for this study. Eight patients were excluded from the study due to initial assessments revealing conditions falling under exclusion criteria (1 patient lacked a prior diagnosis with a COVID-19 infection swab, 2 had concurrent tumor pathologies, 3 exhibited systemic inflammation, and 2 had skin infections), and 23 patients chose to undergo a rehabilitation program at a rehabilitative gym instead. Participants were randomly assigned to one of two rehabilitation treatment groups: the group treated at a health resort facility (Group A, n=36) and the group performing the exercise program at home (Group B, n=36). However, 6 patients did not complete follow-up assessments at different time points, resulting in the final evaluation of data collected from 66 patients, with 33 allocated to Group A and 33 to Group B (Fig. 1).

The patient enrollment was conducted between January 2023 and April 2023. Patients in group A underwent a 5-week rehabilitation cycle with two weekly sessions, totaling 10 sessions, in a health resort setting. The patients underwent treatments at two health resort facilities located in the Euganean Basin, Veneto, Italy, equipped with pools of the same depth, size, and water type. Patients in group B underwent a 5-week rehabilitation cycle at home with two weekly sessions, totaling 10 sessions.

At the beginning (T0) and at the end (T1) of the treatment, and during two subsequent follow-up times at 3 months (T2) and 6 months (T3), after the end of the treatment, patients in both groups were evaluated.

ELIGIBILITY:
The inclusion criteria for the study included the following requirements: age between 18 and 75 years; a previous COVID-19 infection occurring between 6 and 18 months before our initial assessment; negative results in tests for the nucleic acid of the SARS-CoV-2 virus conducted on respiratory samples, such as oropharyngeal swabs; body temperature ≤ 37°C; presence of reduced cardio-respiratory capacity and/or motor deficits caused by the SARS-CoV-2 virus infection; manifestation of possible cognitive symptoms that could not be attributed to other conditions; no participation in cycles of thermal mineral-rich therapy in the six months preceding the study.

Exclusion criteria from the study included: inability to understand and sign the informed consent form; absence of a previous positive detection of nucleic acid of the SARS-CoV-2 virus in tests on respiratory samples; current positivity for the nucleic acid of the SARS-CoV-2 virus in respiratory samples; epilepsy, severe psychiatric disorders, neoplasms, or pregnancy. Moreover, commonly recognized contraindications for health resort treatments, such as skin infections or open wounds, systemic inflammation, heart, liver, respiratory, or kidney failure, and urinary or fecal incontinence, were considered additional exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | immediately before and after intervention and 3 and 6 months follow-ups
  a commonly used pain assessment tool that involves asking patients to rate their pain verbally or visually on a scale from 0 to 10, with 0 indicating no pain and 10 representing the worst possible pain
Hand grip strength | immediately before and after intervention and 3 and 6 months follow-ups
  the strength of the dominant hand was assessed using a digital handheld dynamometer
Barthel Dyspnea Scale | immediately before and after intervention and 3 and 6 months follow-ups
  The Barthel Dyspnea Scale is a validated tool used to measure the severity of dyspnea. It evaluates various activities and tasks that may provoke dyspnea, allowing to assess and monitor the impact of dyspnea on a patient's daily life
Fatigue Assessment Scale | immediately before and after intervention and 3 and 6 months follow-ups
  a self-report questionnaire designed to assess the severity and impact of fatigue. It consists of 10 items, describing different aspects of fatigue.
Beck's Depression Inventory (BDI | immediately before and after intervention and 3 and 6 months follow-ups
  the BDI is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression
Beck Anxiety Inventory (BAI) | immediately before and after intervention and 3 and 6 months follow-ups
  the BAI is a self-report questionnaire designed to assess the severity of anxiety symptoms and consists of 21 items that measure various aspects of anxiety
12-Item Short Form Health Survey (SF-12) | immediately before and after intervention and 3 and 6 months follow-ups
  The SF-12 is employed for assessing health-related quality of life (HRQoL). It is a shortened version of the SF-36, consisting of 12 items that measure eight health domains, including physical functioning, limitations due to physical health problems, bodily pain, general health perception, vitality, social functioning, limitations due to emotional problems, and mental health

SECONDARY OUTCOMES:
Patients satisfaction | immediately after intervention
  Specifically designed questionnaire (Likert scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Universityof Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: No